CLINICAL TRIAL: NCT06827470
Title: Open-label, Phase 1/2, Dose-escalation Clinical Trial to Establish a Controlled Human Infection Model by Determining and Confirming the Optimal and Safe J820 Bordetella Pertussis Dose Administered Intranasally to Healthy Adults 18-50 Years of Age That Induces Mild Symptomatic Infection and Detection of B. Pertussis in Nasal Samples
Brief Title: Establishing a Controlled Human Infection Model of Pertactin-deficient Bordetella Pertussis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CD2301; 75D30123C17596 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC))
Record Dates: First submitted 2025-01-14; First posted 2025-02-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pertussis (Whooping Cough)
Keywords: Bordetella pertussis; Pertussis; Whooping cough; Controlled human infection model; Human challenge; Phase 1 clinical trial; Immune response
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Dose Number 5 (10^5) (Experimental)
  Interventions: Biological: Biological: Bordetella pertussis J820
- Group 2: Dose Number 7 (10^6) (Experimental)
  Interventions: Biological: Biological: Bordetella pertussis J820
- Group 3: Dose Number 9 (10^7) (Experimental)
  Interventions: Biological: Biological: Bordetella pertussis J820
- Group 4: Dose Number 11 (10^8) (Experimental)
  Interventions: Biological: Biological: Bordetella pertussis J820
- Group 5: Dose Number 13 (10^9) (Experimental)
  Interventions: Biological: Biological: Bordetella pertussis J820

INTERVENTIONS:
Biological: Biological: Bordetella pertussis J820 — Intranasal inoculation of Bordetella pertussis J820 in each naris on Day 1 of the study.

SUMMARY:
The overall goal of this study is to establish a PRN-deficient pertussis Controlled Human Infection Model (CHIM) that represents currently circulating isolates, in the context of a North American exposure (vaccination and infection) pedigree.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy ALL of the following criteria:

1. Age 18-50 years, inclusive.
2. Good general health status, as determined by history and physical examination conducted no longer than 30 days prior to the challenge.
3. Participants who, in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g., complete Diary Cards, return for follow-up visits).
4. Written informed consent obtained from the participant.
5. If a cis woman and/or gender divergent person is at risk of becoming pregnant has practiced adequate contraception for 28 days prior to challenge and has a negative pregnancy test on the day before B. pertussis challenge and has agreed to continue adequate contraception until 60 days after inoculation.

Risk of pregnancy is defined as any individual assigned female at birth or with reproductive capacity who is sexually active with individuals with sperm-producing capabilities. Individuals who have received the following are considered to not have reproductive capacity:

* Documented hysterectomy
* Documented bilateral salpingectomy
* Documented bilateral oophorectomy
* Documented and current bilateral tubal ligation or occlusion
* Credible self-reported history of diagnosed infertility
* Hormone therapy (e.g., testosterone), provided it is administered consistently and medically assessed as sufficient to reduce pregnancy such that ovulation has ceased
* Any other condition, as determined by the Principal Investigator, that would render an individual incapable of becoming pregnant

Adequate contraception is defined as a contraceptive method with a failure rate of <1% per year when used consistently and correctly and, when applicable, in accordance with the product label. Examples include the following:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable
* Intra-uterine device (IUD) with or without hormonal release
* Vasectomized partner, if this is the participant's sole partner and the partner has received a medical assessment of the surgical success
* Credible self-reported history of abstinence for at least 28 days prior to challenge

Exclusion Criteria:

Participants with ANY of the following criteria at the time of screening will be excluded:

1. Underlying chronic medical condition requiring ongoing follow-up and monitoring by a physician (e.g., diabetes, seizure disorder).
2. Underlying cardiac and/or pulmonary disease including hypertension, angina, prior myocardial infarction, asthma, emphysema, chronic bronchitis, and pulmonary tuberculosis.
3. Moderate or severe symptoms of health anxiety, anxiety, and mood symptoms. Self-reported current diagnosis of a major psychiatric illness, including a schizophrenia spectrum disorder, bipolar disorder, posttraumatic stress disorder, obsessive compulsive disorder, substance use, or eating disorder.
4. QT prolongation on electrocardiogram (EKG).
5. History of everyday smoking/vaping in the last 2 years and/or current smoking/vaping more than once per week.
6. Pregnant (known before or established at the time of screening using a urine-based test) or breastfeeding.
7. Immunocompromised (with HIV/AIDS-positive or receiving immunosuppressive therapy involving steroids) or with any medical condition or medication that leads to a compromised immune system.
8. Positive for hepatitis B or C by blood test.
9. Vaccinated against pertussis within previous 5 years and/or >7 cumulative doses from infancy to date of screening.
10. Reported history of laboratory-confirmed pertussis infection, including having been exposed to B. pertussis in a Controlled Human Infection Model
11. Antibody titer to pertussis toxin >20 IU/mL (2x the lower limit of quantification (LLOQ)).
12. Detection of B. pertussis in nasal samples prior to challenge using culture isolation and/or PCR detection, or detection of other respiratory infection.
13. Living or working with (any form of close contact) any of the at-risk/vulnerable groups who are not up to date on their vaccination, specifically children <1 year of age, pregnant woman who have not yet received their maternal Tdap vaccine, immunocompromised individuals, adults >65 years of age who have not received a dose of Tdap vaccine within the past 10 years, or other at risk persons, as applicable, up to Day 57.

    Note: Household members whose vaccination is not current will be offered or directed to a pertussis-containing vaccine, as recommended and funded by the Nova Scotia Department of Health and Wellness.
14. Known allergy to macrolides including azithromycin or erythromycin, history of Clostridium difficile within last 2 months.
15. Any contraindication to receiving azithromycin.
16. Taking any systemic antibiotic currently or within the previous 2 weeks.
17. Currently taking terfenadine, astemizole, theophylline, or cimetidine.
18. Poor venous access, as defined by inability to obtain venous blood after 3 venipuncture attempts.
19. Recent (within 6 months) nasal or sinus surgery, recent use of intranasal steroids (4 weeks), or diagnosis with nasal polyps.
20. Receipt of any investigational drug or vaccine within 6 months prior to challenge. An investigational vaccine is defined as a vaccine that is still being tested in clinical trials or one that has not yet been authorized for use in Canada for administration by public vaccine programs.
21. Receipt of any authorized vaccines within 2 weeks prior to challenge with B. pertussis in this study. (This is to avoid attributing any AEs from these vaccines to the B. pertussis challenge, which would skew the study results.)
22. Previous moderate or severe respiratory infection that required hospitalization.
23. Head trauma (e.g., fracture of the cribriform plate) within 1 year of screening.
24. Any other finding that the Investigator considers will make the participant unsuitable for the study or unable to comply with the study requirements.
25. Symptoms indicative of acute respiratory illness (such as fever, cough, difficulty breathing) identified during the physical examination done on Day -1 (check-in) or Study Day 1 before a participant is challenged.
26. History of Bell's Palsy and/or facial paralysis.
27. Receipt of facial cosmetic filler in the past 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures | Study Day 1 up to Study Day 29
  Establish a PRN-deficient pertussis CHIM that identifies the lowest challenge dose that successfully & safely infects nearly all (≥85%) participants challenged (HID) & produces the highest achievable rate of symptomatic infection (HSD), including cough, using an adaptive dose response design.
  This is contingent upon determining each participant's clinical outcome post-challenge to compute the rate of symptomatic infection & rate of overall infection per dose group, based on outcomes for all participants receiving that dose. As a derived variable, clinical outcomes will be measured/determined using programmed case definitions previously designed to emulate the natural course of early pertussis disease following experimentally induced pertussis infection. Clinical outcome measures include:
  1. B. pertussis lab testing of samples (culture, PCR, serology)
  2. Clinical assessments (safety bloods, physical exams, DCs, symptom self-reporting).

SECONDARY OUTCOMES:
Secondary Outcome Measures | Study Day 1 up to Study Day 29
  • To measure the rate of cough and describe the clinical presentation via:
  1. Self-reporting
  2. Clinical assessment
Secondary Outcome Measures | Day 1 up to Study Day 181
  • To evaluate the immune response following challenge associated with infection via:
  1. Humoral immune responses (analyte; unit; sample; technique):
  A) Anti-PT Antibodies; IU/mL; Serum; ELISA B) Anti-FHA Antibodies; IU/mL; Serum; ELISA C) Anti-PRN Antibodies; IU/mL; Serum; ELISA D) Anti-FIM Antibodies; EU/mL; Serum; ELISA
Secondary Outcome Measure | Time Frame: Day 1 up to Study Day 181
  • To evaluate the immune response following challenge associated with infection via:
  2. Cellular & Cellular-mediated immune responses
  Cellular:
  A) Eotaxin-2, Perfornin, Granzyme-A & Granzyme-B; all pg/mL, by nasal wash using Luminex
  Cellular-mediated:
  A) Neutrophil CD16+, B cell CD19+, T Cell CD4+, T cells CD8+, Mucosal associated invariant T cell(MAIT) cells, NK cell CD3-CD56+, Monocyte CD14+, Eosinophil Siglec8+, gamma delta T cell; all % & absolute count, by whole blood & nasal swab using Flow cytometry
Secondary Outcome Measures | Study Day 1 up to Study Day 29
  • To explore the time course of azithromycin therapy in clearing infection and/or symptoms, via testing during treatment as applicable via:
  1. B. pertussis laboratory testing of samples (culture, PCR): A) The mean number of days to culture negativity (i.e., bacterial count of zero in both NW and NPA samples) in days (with a 95% confidence interval) following treatment.
  B) The mean number of days to PCR negativity (i.e., PCR negative for each of the targets, that is IS481 and ptxS1 in both NW and NPA samples in days (with a 95% CI) following treatment.
  C) The cumulative proportion of participants that are negative by day following treatment by culture and PCR.
Secondary Outcome Measure | Time Frame: Study Day 1 up to Study Day 29
  • To explore the time course of azithromycin therapy in clearing infection and/or symptoms, via testing during treatment as applicable via:
  2. Clinical assessments (as needed): A) The mean number of days to symptom resolution (i.e., no reporting/detection of symptoms and/or signs) in days (with a 95% confidence interval) following treatment.
  B) The cumulative proportion of participants with resolved pertussis symptoms by day following treatment.

OTHER OUTCOMES:
Exploratory Outcome Measures | Study Day 1 up to Study Day 181
  • To recommend optimal time points for the collection of biological specimens that facilitate studying mucosal and systemic immune responses to pertussis infection and/or vaccination will be measured via:
  1. Collective review of the results from all laboratory testing conducted to measure the previous outcomes.
Exploratory Outcome Measures | Study Day 1 Up to Study Day 181
  • Contributing samples from the study to the CDC biorepository will be measured via:
  1. Estimating the proportion of samples for which a portion will be submitted to the biorepository.

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Center for Vaccinology, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No